CLINICAL TRIAL: NCT04420338
Title: SeroCOVIDial Study: Assessment of SARS-COV2 Seroconversion in Patients on Chronic Hemodialysis and in Their Caregivers, a Cohort Study
Brief Title: SeroCOVIDial Study: Assessment of COVID-19 Seroconversion in Patients on Chronic Hemodialysis and in Their Caregivers, a Cohort Study
Acronym: SeroCOVIDial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-34; 2020-A01515-34 (Registry Identifier: ID RCB)
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Chronic Hemodialysis Patients; Caregivers of Chronic Hemodialysis Patients
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic hemodialysis patients (Experimental)
  Interventions: Biological: Blood sample; Biological: Serum tube collection
- Caregivers of chronic hemodialysis patients (Experimental)
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — rapid serological tests carried out
Biological: Serum tube collection — SARS-COV2 seroconversion assay
  Arms: Chronic hemodialysis patients

SUMMARY:
Background: The preventive containment measures implemented in the COVID-19 pandemic are not feasible in chronic hemodialysis patients (HD) who need to attend their dialysis sessions 3 times a week. HD patients display frequent comorbidities (such as diabetes and cardiovascular disease), and immune deficiency, which expose them to an increased risk of severe forms of COVID-19. They can be infected in their dialysis center despite the measures taken to limit this risk. Their caregivers are also at risk of infection if patients carry the virus. Dialysis centers face major organizational challenges in terms of patient and caregiver safety. Knowing the viral serological status of HD patients and caregivers, the proportion of asymptomatic forms, and the persistence and effectiveness of immunization over time would be of major interest for patient management and the organization of dialysis care.

Research objectives: The primary objective of SeroCOVIDial is to assess the prevalence of SARS-COV2 seroconversion at inclusion (M0) in a cohort of HD patients, using the rapid serological test. Secondary Objectives : 1) assess the prevalence of SARS-COV2 seroconversion in dialysis caregivers at M0, using the same test; 2) assess the proportion of asymptomatic forms of COVID-19 in HD patients and in their caregivers; 3) compare the prevalence of seroconversion and the proportion of asymptomatic forms in HD patients according to their clinical characteristics and co-morbidities; 4) assess the prevalence of SARS-COV2 seroconversion in participants who had a documented COVID-19; 5) evaluate the spread of the epidemic and the kinetics of seroconversion in patients and caregivers by a second test performed at M3; 6) evaluate the predictive value of SARS-COV2 seroconversion at M0 on the risk of developing a symptomatic COVID-19 infection within 6 months, in patients and caregivers; 7) evaluate a posteriori the intrinsic diagnostic performances of the test in comparison with serological gold standards (ELISA and seroneutralization).

Methods: Multicenter cohort study, carried out in 4 dialysis facilities in Aix-Marseille.

Procedure: collection of clinical data and rapid serological tests carried out at M0 and M3, in patients and caregivers (a systematic screening for COVID-19 symptoms has been carried out in all HD patients in the 4 participating centers since the beginning of the pandemic in France).

Number of participants: 800 eligible persons (561 HD patients, and 239 caregivers). Material tested: rapid Biosynex serological test on 1 drop of blood, and 1 tube of frozen serum for patients at M0 and M3. Clinical data will also be collected.

Primary endpoint: prevalence of SARS-COV2 seroconversion in HD patients. Maximum duration of participation for each patient: 6 months. Duration of research: 6 months and 2 weeks (inclusions over 2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Subject of 18 years of age or older
* Chronic hemodialysis patients or caregiver of chronic hemodialysis patients
* signed consent
* Social Security affiliation.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Minors
* Adults under guardianship and trusteeship, persons deprived of their liberty,
* Participation in a SARS-COV2 vaccine study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
The prevalence of SARS-COV2 seroconversion in chronic hemodialysis patients | 6 months
  Proportion of positive patients out of the total number of patients tested

SECONDARY OUTCOMES:
The prevalence of SARS-COV2 seroconversion in dialysis caregivers | 6 months
  Proportion of positive caregivers out of the total number of caregivers tested

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARBAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, PACA, France

IPD SHARING:
Plan to Share IPD: No